CLINICAL TRIAL: NCT01288287
Title: A Prospective, Multicentre, Non-interventional, Observational, Cohort Study to Evaluate the Long Term Clinical, Patient Reported and Health Care Resource Utilization Effects of an Early Response to Certolizumab Pegol (Cimzia®) in Rheumatoid Arthritis Patients in Daily Clinical Practice in the United Kingdom and Eire.
Brief Title: Long Term Effects of an Early Response to Certolizumab Pegol (CZP, Cimzia®) in Rheumatoid Arthritis (RA) Patients
Acronym: RA-PROACTIVE
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: RA0042
Record Dates: First submitted 2011-01-25; First posted 2011-02-02 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-08

CONDITIONS: Arthritis,Rheumatoid
Keywords: Certolizumab pegol; Cimzia®
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Week 12 Disease Activity Score (DAS) Responders: Patients achieving a reduction from Baseline in a Disease Activity Score 28-joint count (Erythrocyte Sedimentation Rate) [DAS28(ESR)] score of greater than 1.2 points at Week 12
- Week 12 Disease Activity Score (DAS) Non-Responders: Patients who fail to achieve a reduction from Baseline in a Disease Activity Score 28-joint count (Erythrocyte Sedimentation Rate) [DAS28(ESR)] score of greater than 1.2 points at Week 12

SUMMARY:
To determine if early clinical response at 12 weeks to Certolizumab Pegol (CZP, Cimzia ®) therapy in adult Rheumatoid Arthritis (RA) patients is a predictor of better long term clinical response at 18 months compared with a lack of clinical response at 12 weeks.

DETAILED DESCRIPTION:
Clinical response will be assessed by the percentage of patients achieving a reduction from Baseline in Disease Activity Score 28-joint count (Erythrocyte Sedimentation Rate) [DAS28(ESR)] score of greater than 1.2 points, which is considered the minimum clinically important difference.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is signed and dated
* The patient is considered capable of and prepared to adhere to the study protocol procedures
* The patient is prescribed CZP according to the Summary of Product Characteristics (SmPC) (UK and Eire) and National Institute of Clinical Excellence (NICE) (UK only) guidelines for anti tumor necrosis factor (TNF) α therapy for Rheumatoid Arthritis (RA).
* The patient is screen-negative for tuberculosis
* The patient is 18 years of age or above

Exclusion Criteria:

* The patient has been exposed previously to biological disease modifying anti rheumatic drugs (DMARD) agents.
* Patient has previously participated in this study or the patient has previously been assigned to treatment in a study of CZP or another biological agent used to treat RA.
* Patient has participated in another study within the last 30 days
* Patient has any medical or psychiatric condition that, in the opinion of the physician, can jeopardize or would compromise the patient's ability to adequately participate in the study
* Patient has inadequate literacy to understand and complete the questionnaires.
* Contraindications stated in the SmPC
* Patient is pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient presenting with Rheumatoid Arthritis (RA) and having prescribed certolizumab pegol (CZP, Cimzia®) at the clinic
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2011-07; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (22):
- 2, Cork, Cork, Ireland
- United Kingdom (21):
  - 7, Bridgend, Bridgend
  - 25, Cardiff, Cardiff
  - 4, Durham, County Durham
  - 17, Poole, Dorset
  - 24, Eastbourne, East Sussex
  - 13, Southend, Essex
  - 11, Manchester, Greater Manchester
  - 12, Manchester, Greater Manchester
  - 6, Southampton, Hampshire
  - 20, Gillingham, Kent
  - 15, St Helens, Lancashire
  - 10, Liverpool, Merseyside
  - 22, Ashford, Middlesex
  - 14, Abergavenny, Monmouthshire
  - 5, Bath, Somerset
  - 19, Burton, Staffordshire
  - 3, Chertsey, Surrey
  - 18, Birmingham, West Midlands
  - 16, Cannock, West Midlands
  - 9, Dudley, West Midlands
  - 1, York, Yorkshire

REFERENCES:
- [Derived] Kumar N, Naz S, Quinn M, Ryan J, Kumke T, Sheeran T. Treatment of Rheumatoid Arthritis with Certolizumab Pegol: Results from PROACTIVE, a Non-Interventional Study in the UK and Ireland. Adv Ther. 2018 Sep;35(9):1426-1437. doi: 10.1007/s12325-018-0758-1. Epub 2018 Aug 3. PMID 30076523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study started to enroll patients in July 2011 in the United Kingdom and Ireland.
Pre-assignment Details: Of the 149 enrolled patients, 147 are included in the Safety Set.
Groups:
- All Patients: Patient presenting with Rheumatoid Arthritis (RA) and having prescribed certolizumab pegol (CZP, Cimzia®) at the clinic.
Period: Overall Study
Arm/Group | All Patients
Started | 149
Safety Set | 147
Full Analysis Set | 111
Completed | 103
Not Completed | 46
Not completed — Lost to Follow-up | 8
Not completed — Withdrawal by Subject | 4
Not completed — Lack of Efficacy | 13
Not completed — Other Reason | 13
Not completed — Unknown Reason | 1
Not completed — Unknown Status | 7

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to the Safety Set, consisting of all patients entered into the study who took at least one dose of Certolizumab Pegol.
Groups:
- Safety Set (All Patients): Patient presenting with Rheumatoid Arthritis (RA) and having prescribed certolizumab pegol (CZP, Cimzia®) at the clinic.
  Safety Set consists of all patients entered into the study who took at least one dose of Certolizumab Pegol.
Arm/Group | Safety Set (All Patients)
Number analyzed (Participants) | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (11.85)
Age, Customized [Number; unit: participants]
  < 65 years | 111
  >= 65 years | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Disease Activity Score (DAS) Response at 78 Weeks Where DAS Response is Defined as a Reduction From Baseline in DAS 28-joint Count (Erythrocyte Sedimentation Rate) [DAS28(ESR)] Score of Greater Than 1.2 Points
Description: DAS28(ESR) is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC), ESR (mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm). 28 joints are examined using:
  DAS28(ESR) = 0.56 * √(TJC) + 0.28* √(SJC) + 0.70* ln(ESR) + 0.014* PtGADA, with TJC=0 to 28, SJC=0 to 28, PtGADA=0 to 100 mm, ESR=0 to infinite mm/hour but ESR values of greater 250 mm/h are typically measurement errors.
  DAS28(ESR) ranges from 0 to around 10 with lower scores indicating less disease activity.
Time Frame: Baseline (Week 0), 78 weeks
Population: Full Analysis Set (FAS) consists of all patients entered into the study who take at least one dose of Certolizumab Pegol and have a valid, non-missing complete DAS28(ESR) score at Baseline and Week 12 (+/- 2 weeks).
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Week 12 Disease Activity Score (DAS) Responders | Week 12 Disease Activity Score (DAS) Non-Responders
Number analyzed (Participants) | 44 | 14
percentage of patients | 79.5 [64.7 to 90.2] | 50.0 [23.0 to 77.0]

2. Secondary Outcome: Change From Baseline in Disease Activity Score 28-joint Count (Erythrocyte Sedimentation Rate) [DAS28(ESR)] Score at 78 Weeks
Description: as for outcome 1
Time Frame: Baseline (Week 0), 78 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Week 12 Disease Activity Score (DAS) Responders | Week 12 Disease Activity Score (DAS) Non-Responders
Number analyzed (Participants) | 44 | 14
units on a scale | -2.45 (1.454) | -1.63 (1.157)

3. Secondary Outcome: Percentage of Participants With a Disease Activity Score (DAS)-Based European League Against Rheumatoid Arthritis (EULAR) Response at 78 Weeks Compared to Baseline
Description: Percentage of patients achieving good, moderate, or no EULAR clinical response, where good response is defined as DAS28(ESR) ≤ 3.2 and decrease from baseline by > 1.2; moderate response is defined as achievement of one of the following:
  * DAS28(ESR) ≤ 3.2 and decrease from baseline > 0.6 and ≤ 1.2,
  * DAS28(ESR) > 3.2 and ≤ 5.1 and decrease from baseline > 0.6,
  * DAS28(ESR) > 5.1 and decrease from baseline > 1.2 Patients without a good or moderate response are considered to be non-responders.
Time Frame: Baseline (Week 0), 78 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Week 12 Disease Activity Score (DAS) Responders | Week 12 Disease Activity Score (DAS) Non-Responders
Number analyzed (Participants) | 44 | 14
percentage of patients
  Good Response | 47.7 | 35.7
  Moderate Response | 36.4 | 50.0
  No Response | 15.9 | 14.3

4. Secondary Outcome: Change From Baseline in Rheumatoid Arthritis Disease Activity Index (RADAI) Scores at 78 Weeks
Description: RADAI is a five-item questionnaire administered to patients. The final score range is 0-10, with higher scores denoting a worse disease state.
  A negative value in RADAI change from Baseline indicates an improvement from Baseline to 78 weeks.
Time Frame: Baseline (Week 0), 78 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Week 12 Disease Activity Score (DAS) Responders | Week 12 Disease Activity Score (DAS) Non-Responders
Number analyzed (Participants) | 51 | 17
units on a scale | -2.64 (2.262) | -1.78 (3.048)

5. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disease Index (HAQ-DI) Scores at 78 Weeks
Description: HAQ-DI is a questionnaire which measures function and health-related quality of life. The final score range is 0-3, with higher scores denoting greater disability. A negative value in HAQ-DI change from Baseline indicates an improvement from Baseline to 78 weeks.
Time Frame: Baseline (Week 0), 78 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Week 12 Disease Activity Score (DAS) Responders | Week 12 Disease Activity Score (DAS) Non-Responders
Number analyzed (Participants) | 50 | 17
units on a scale | -0.43 (0.506) | -0.34 (0.606)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse drug reactions (TEADRs) were collected up to 88 weeks. TEADRs are events with an onset date from the first dose of Certolizumab Pegol (CZP) to 10 weeks after the last dose of CZP.
Description: Adverse Drug Reactions presented below refer to the Safety Set, consisting of all patients entered into the study who took at least one dose of Certolizumab Pegol.
Arm/Group | Safety Set (All Patients)
Serious Adverse Events (participants affected / at risk) | 8/147
Other Adverse Events (participants affected / at risk) | 3/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Set (All Patients) (N=147)
Cellulitis (Infections and infestations) | 1 (1)
Pulmonary Tuberculosis (Infections and infestations) | 2 (2)
Abortion induced (Surgical and medical procedures) | 2 (2)
Liver function test abnormal (Investigations) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Set (All Patients) (N=147)
Exposure during pregnancy (Injury, poisoning and procedural complications) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days